CLINICAL TRIAL: NCT01243138
Title: Prevalence of Cardiovascular Risk Factors in Patients Attending General Practice Clinics in Selected Countries in the Africa and The Middle East Region
Brief Title: Africa and Middle East Cardiovascular Epidemiological Study
Acronym: ACE
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A2581186
Record Dates: First submitted 2010-11-12; First posted 2010-11-18 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Obesity; Smoking; Dyslipidemia; Diabetes Mellitus; Hypertension
Keywords: Cross-sectional; epidemiological study; to evaluate the prevalence of CV risk factors in patients attending general practice in AfME region
MeSH Terms: conditions — Obesity; Smoking; Dyslipidemias; Diabetes Mellitus; Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Whole Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a cross-sectional, epidemiological study to determine the prevalence of cardiovascular risk factors such as obesity, smoking, dyslipidemia, diabetes mellitus and hypertension in patients attending General Practice clinics in the Africa and Middle East region. A total of 4300 patients will be evaluated. In patients who are found to have previously been diagnosed with cardiovascular (CV) risk factors such as dyslipidemia or hypertension, the level of control of their respective conditions will also be evaluated.

DETAILED DESCRIPTION:
This is a cross-sectional, epidemiological study. In the course of this study, 4,300 persons from general practice, and other non specialist clinics of selected countries of the Africa and Middle East region, will be evaluated for the presence of cardiovascular (CV) risk factors such as obesity, smoking, dyslipidaemia, diabetes mellitus and hypertension. The degree of control of hypertension and dyslipidaemia in those previously diagnosed with these conditions will also be assessed. All medications used for CV risk factor control will also be ascertained.

Patient evaluation will be done by physicians in charge of the selected clinics (who will be trained for case report forms completion) over one visit, through history taking, clinical examination as well as laboratory investigations. Every fifth patient seen on a particular day, fulfilling the inclusion and exclusion criteria would be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 18 or above

Exclusion Criteria:

* Pregnant women and/or lactating mothers
* Subjects presenting with any life threatening disease/condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subject selection would be from clinics in a primary care setting
Sampling Method: Probability Sample
Enrollment: 4386 (Actual)
Dates: Start 2011-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Prevalence of cardiovascular (CV) risk factors such as obesity, smoking, dyslipidemia, diabetes mellitus and hypertension | At the time of the first visit

SECONDARY OUTCOMES:
Compare the prevalence of cardiovascular (CV) risk factors such as obesity, smoking, dyslipidaemia, diabetes mellitus and hypertension in the urban and rural population. | At the time of the first visit
Compare the prevalence of CV risk factors such as obesity, smoking, dyslipidaemia, diabetes mellitus and hypertension in the male and female population. | At the time of the first visit
Stratifying the prevalence of CV risk factors such as obesity, smoking, dyslipidaemia, diabetes mellitus and hypertension by age groups. | At the time of the first visit
Ascertain the level of blood pressure and lipids' control as per the European Society of Cardiology (ESC) guidelines in patients who have been previously diagnosed as hypertensive or dyslipidaemic. | At the time of the first visit
Ascertain the most commonly used medications in those that have been previously diagnosed as diabetic, hypertensive or dyslipidaemic. | At the time of the first visit

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (72):
- Algeria (9):
  - Pfizer Investigational Site, Algiers
  - Pfizer Investigational Site, Bejaja
  - Pfizer Investigational Site, Djelfa
  - Pfizer Investigational Site, Laghouat
  - Pfizer Investigational Site, M'Sila
  - Pfizer Investigational Site, Relizane
  - Pfizer Investigational Site, Saïda
  - Pfizer Investigational Site, Tébessa
  - Pfizer Investigational Site, Tlemcen
- Cameroon (6):
  - Pfizer Investigational Site, Yaoundé, Cite Verte
  - Pfizer Investigational Site, Douala, Deido
  - Pfizer Investigational Site, Bafoussam
  - Pfizer Investigational Site, Mbandjok
  - Pfizer Investigational Site, Njombé
  - Pfizer Investigational Site, Okoa
- Egypt (4):
  - Pfizer Investigational Site, Alexandria
  - Pfizer Investigational Site, Cairo
  - Pfizer Investigational Site, Shiben Al Kom
  - Pfizer Investigational Site, Tanta
- Ghana (5):
  - Pfizer Investigational Site, Accra
  - Pfizer Investigational Site, Jachie-Ashanti
  - Pfizer Investigational Site, Kumasi
  - Pfizer Investigational Site, Sogakope V/R
  - Pfizer Investigational Site, Takoradze
- Jordan (3):
  - Pfizer Investigational Site, Amman
  - Pfizer Investigational Site, Irbid
  - Pfizer Investigational Site, Salt
- Kenya (2):
  - Pfizer Investigational Site, Chongoria
  - Pfizer Investigational Site, Nairobi
- Kuwait (6):
  - Pfizer Investigational Site, Adailiya
  - Pfizer Investigational Site, Al Faḩāḩīl
  - Pfizer Investigational Site, Kuwait City
  - Pfizer Investigational Site, Mishrif
  - Pfizer Investigational Site, Qadesya
  - Pfizer Investigational Site, Yarmouk
- Lebanon (4):
  - Pfizer Investigational Site, Jbeil, Lebanon, Lebanon
  - Pfizer Investigational Site, Beirut
  - Pfizer Investigational Site, Jounieh
  - Pfizer Investigational Site, Tripoli
- Nigeria (5):
  - Pfizer Investigational Site, Abuja, FCT
  - Pfizer Investigational Site, Abuja, Garki
  - Pfizer Investigational Site, Calabar
  - Pfizer Investigational Site, Enugu
  - Pfizer Investigational Site, Keffi, Nassarawa
- Saudi Arabia (5):
  - Pfizer Investigational Site, Dammam
  - Pfizer Investigational Site, Jeddah
  - Pfizer Investigational Site, Mecca
  - Pfizer Investigational Site, Riyadh
  - Pfizer Investigational Site, Yanbu
- Senegal (6):
  - Pfizer Investigational Site, Dakar, Nabil Choucair
  - Pfizer Investigational Site, Dakar, Ouakam
  - Pfizer Investigational Site, Kedoungou
  - Pfizer Investigational Site, Kébémer
  - Pfizer Investigational Site, Saint-Louis
  - Pfizer Investigational Site, Ziguinchor
- South Africa (7):
  - Pfizer Investigational Site, Halfway House, Gauteng
  - Pfizer Investigational Site, Sydenham, Durban, KwaZulu-Natal
  - Pfizer Investigational Site, Mokopane, Limpopo
  - Pfizer Investigational Site, Sheshego, Limpopo
  - Pfizer Investigational Site, Mamelodi East, Pretoria
  - Pfizer Investigational Site, Kwa-Zulu Natal
  - Pfizer Investigational Site, Rondebosch
- Tunisia (6):
  - Pfizer Investigational Site, Aryanah
  - Pfizer Investigational Site, Bouficha
  - Pfizer Investigational Site, Messaadine
  - Pfizer Investigational Site, Sfax
  - Pfizer Investigational Site, Tunis
  - Pfizer Investigational Site, Zaghouan
- United Arab Emirates (4):
  - Pfizer Investigational Site, Abu Dhabi
  - Pfizer Investigational Site, Al Ain City
  - Pfizer Investigational Site, Dubai
  - Pfizer Investigational Site, Ras Al Khaima

REFERENCES:
- [Derived] Hamoui O, Omar MI, Raal FJ, Rashed W, Kane A, Alami M, Abreu P, Mashhoud W, Alsheikh-Ali AA. Increases in statin eligibility to reduce cardiovascular risk according to the 2013 ACC/AHA cholesterol guidelines in the Africa Middle East region: a sub-analysis of the Africa Middle East Cardiovascular Epidemiological (ACE) study. BMC Cardiovasc Disord. 2019 Mar 15;19(1):61. doi: 10.1186/s12872-019-1034-2. PMID 30876390
- [Derived] Brouri M, Ouadahi N, Nibouche D, Benabbas Y, El Hassar M, Bouraoui S, Abad N, Abreu PC, Ikardouchene L. [Cardiovascular risk factors in Algeria. Analysis of the subgroup from the "Africa/Middle East Cardiovascular Epidemiological" Study]. Ann Cardiol Angeiol (Paris). 2018 Apr;67(2):61-66. doi: 10.1016/j.ancard.2018.01.003. Epub 2018 Mar 9. French. PMID 29530274
- [Derived] Raal FJ, Alsheikh-Ali AA, Omar MI, Rashed W, Hamoui O, Kane A, Alami M, Abreu P, Mashhoud WM. Cardiovascular risk factor burden in Africa and the Middle East across country income categories: a post hoc analysis of the cross-sectional Africa Middle East Cardiovascular Epidemiological (ACE) study. Arch Public Health. 2018 Feb 12;76:15. doi: 10.1186/s13690-018-0257-5. eCollection 2018. PMID 29449941
- [Derived] Ahmed AM, Hersi A, Mashhoud W, Arafah MR, Abreu PC, Al Rowaily MA, Al-Mallah MH. Cardiovascular risk factors burden in Saudi Arabia: The Africa Middle East Cardiovascular Epidemiological (ACE) study. J Saudi Heart Assoc. 2017 Oct;29(4):235-243. doi: 10.1016/j.jsha.2017.03.004. Epub 2017 Mar 14. PMID 28983166
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2581186&StudyName=Africa%20and%20Middle%20East%20Cardiovascular%20Epidemiological%20Study